CLINICAL TRIAL: NCT00225199
Title: A Multicenter, Double-blind, Randomized, Placebo-controlled, Parallel-group Study to Investigate the Efficacy and Safety of Daily Oral Administration of SH T00660AA for the Treatment of Endometriosis Over 12 Weeks
Brief Title: Efficacy and Safety of SH T00660AA in Treatment of Endometriosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Therapeutic Area Head, Bayer Schering Pharma AG
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 91233; 307041
Record Dates: First submitted 2005-09-22; First posted 2005-09-23 (Estimated); Last update posted 2010-04-23 (Estimated); Status verified 2010-04

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Visanne (BAY86-5258, SH T00660AA)
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Visanne (BAY86-5258, SH T00660AA) — orally once daily
  Arms: Arm 1
Drug: Placebo — orally once daily
  Arms: Arm 2

SUMMARY:
The purpose of this study is to demonstrate safety and efficacy of SH T00660AA compared to placebo in the treatment of endometriosis

DETAILED DESCRIPTION:
The study has previously been posted by Schering AG, Germany. Schering AG, Germany has been renamed to Bayer Schering Pharma AG, Germany.

Bayer Schering Pharma AG, Germany is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with endometriosis-associated pelvic pain

Exclusion Criteria:

* Pregnant or lactating women
* history or suspicion of hormone dependent tumor
* therapy resistant endometriosis
* need for primary surgical treatment
* any other conditions which forbid the participation.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 198 (Actual)
Dates: Start 2004-03; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Efficacy | Assessment of pain relief at end of treatment

SECONDARY OUTCOMES:
Adverse event collection | Assessment at end of study
Treatment satisfaction by patient | Assessment at end of study

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer

REFERENCES:
- [Derived] Sieverding M, Gerlinger C, Seitz C. Substituting a randomised placebo control group with a historical placebo control in an endometriosis pain trial: a case study re-evaluating trial data using historical control data from another trial. BMJ Open. 2023 Jul 21;13(7):e063188. doi: 10.1136/bmjopen-2022-063188. PMID 37479520